CLINICAL TRIAL: NCT02932111
Title: Effectiveness of Osteopathic Manipulative Therapy for Managing Symptoms of Irritable Bowel Syndrome. A Prospective Randomized Study -IBSOMT
Brief Title: Irritable Bowel Syndrome and Osteopathic Manipulative Therapy
Acronym: IBSOMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150920
Record Dates: First submitted 2016-10-07; First posted 2016-10-13 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Osteopathic manipulative treatment; pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic session (Experimental): The osteopath put fingers on abdominal projection of the junction and sinks deeply into the abdomen until it perceives the trigger zone. Once in contact with the sphincter, it performs friction in the hourly sense, vibration, inhibitions or rebounds.
  Interventions: Procedure: osteopathic session
- Placebo manipulative session (Placebo Comparator): The Osteopath will touch the patient's limbs at the same place of osteopathic manipulative treatment, but without any intention of treatment and without any known and indexed reproduction techniques to simulate an osteopathic treatment, without its benefits.
  Interventions: Procedure: Placebo manipulative session

INTERVENTIONS:
Procedure: osteopathic session — 3 osteopathic manipulative sessions. An six-week double-blind treatment period lasting from week 2 (Visit V1) until week 6, Visit 3.
  Arms: Osteopathic session
Procedure: Placebo manipulative session — 3 osteopathic manipulative sessions. An six-week double-blind treatment period lasting from week 2 (Visit V1) until week 6, Visit 3.
  Arms: Placebo manipulative session

SUMMARY:
The Irritable Bowel Syndrome (IBS) is defined by a combination of abdominal pain, bowel dysfunction during recurrent periods of shorter or longer duration. The absence of well-defined pathophysiological marker requires a clinical definition. The most used are the Rome criteria III whose version was published in 2006 and version IV under development.

An epidemiological study conducted in 2003 in Europe in 8 countries with over 42 000 people, found on the basis of questionnaires a prevalence of 11.5% with a diagnosis of IBS of 4.8%.in the total population; the results of this study were comparable to data obtained in the USA. A French work of our team at 35 447 healthy adults found a 6.2% frequency. In all these studies, there is a very large predominance of women (sex ratio near 2), with a preponderance of subjects of the age group 40-50 years.

IBS economic weight is high, partly due to costs directly incurred by the IBS and the costs generated by associated diseases: number of visits to the general practitioner, to the specialist, the prescription and realization of complementary examinations, hospitalization, purchase drugs and work stoppage.

From a pathophysiologic perspective, IBS is now considered as a multifactorial disease involving varying degrees, depending on the individual variables, visceral hypersensitivity, disturbances of digestive motility, impaired sensorimotor way communications between the gastrointestinal tract and the central nervous system, intestinal micro-inflammation.

Hypothesis of this search is that the osteopathic manipulative treatment (OMT) will improve the symptomatology of IBS in patients with functional gastrointestinal disorders.

DETAILED DESCRIPTION:
The Irritable Bowel Syndrome (IBS) is defined by the association between abdominal pain, bowel dysfunction for longer or shorter periods of time, but in any case, recurring. The absence of well-defined pathophysiological marker, requires a clinical definition. The most used are the Rome criteria III whose version was published in 2006, Version IV is under development.

coordinator's team demonstrated in a randomized, placebo-controlled, 31 patients with refractory IBS, visceral osteopathy that is associated with a significant improvement in diarrhea, abdominal distension and abdominal pain without change constipation. This improvement was associated with a decrease in rectal sensitivity without changes of depression, time of total or segmental colonic transit. This effect persisted one year after the end of this essay.

Primary objective To evaluate the efficacy of osteopathic manipulative treatment on IBS symptoms in IBS adult patients over a 3-sessions period according to our preliminary study (73).

Secondary objectives To evaluate and to compare the results of two therapeutic modalities : osteopathic manipulative treatment and placebo manipulative treatment on

* Subjective clinical criteria: Constipation, Diarrhea, abdominal pain, bloating, topology of abdominal pain.
* Improvement of quality of life
* Decrease of depression and anxiety
* Changes in the medication after treatment
* Search for a possible practitioner effect.

Experimental design:

Double-blind, randomized, placebo-controlled study, parallel group multicenter French study of 3 OMT sessions followed by an 18-week follow-up period.

Patients will be randomized in a 1:1 ratio to receive osteopathic manipulative treatment or placebo manipulative treatment every 2 weeks with stratification according to the IBS phenotype (IBS-C, IBS-D, IBS-M, IBS-U).

Description of research methodology

Design Double blind randomized clinical trial with a distribution of subjects in groups at a ratio (1:1) It is a double blind, multicenter, comparative, prospective, two-arms randomized study.

* One group of patients will benefit from OMT for the treatment of irritable bowel syndrome.
* One group of patients will receive a placebo manipulation therapy for the treatment of irritable bowel syndrome Schedule

The schedule will include 7 visits:

* Four medical visits: V0 (inclusion), V4 (at week 8), V5 at week 12 and V6 at week 24 respectively;
* Three osteopathic visits (V1, V2, V3) that correspond to the visceral or placebo manipulative treatment at week 2, 4, and 6, respectively.
* If patients, are not able to immediately participate to the study a screening visit (VS) could be added in order to separate the decision of participation and the beginning of the study.

Efficacy assessment The main criteria for treatment efficacy are the value of the IBS severity score. The IBS severity score was established from the self-administered questionnaire developed and validated by Francis. The French version was validated by the MAPI Research Institute. This questionnaire includes two items concerning abdominal pain and abdominal bloating (yes/no) and four visual analog scales (1-100) to assess the severity of abdominal pain, bloating, relief after stool, and impact of symptoms on quality of life. The number of days the patient suffered during the last 10 days was also recorded. The responses were used to calculate a quantitative severity score from 0 to 500 used to make a qualitative classification: severity score 75-175 = mild, 175-300 = moderate, > 300 = severe.

This questionnaire will be registered 7 times, at inclusion (V0), during each osteopathic visit (V1, V2, V3) and each medical visit (V4, V5, V6):

* Before treatment at (V0),
* During visceral manipulative treatment (V1, V2, V3)
* During the follow-up period, after visceral manipulative treatment (osteopathic or placebo),

  * At 8 weeks (V4) after inclusion,
  * At 12 weeks (V5) after inclusion and
  * At 24 weeks (V6) at the end of follow up visit In each center, local osteopaths will be learned to provide the same placebo or osteopathic manipulation

Number of subjects chosen: 210 patients Sample Size Considering that the minimal clinical difference on the primary outcome measure that would lead clinicians to change the treatment is 50 points the IBS Symptom Severity Score, and that the standard deviation of this variable is 105 points, the sample size required to detect a difference at 90% power and 5% two-sided significance level is 94 patients/group .

To allow for loss to follow up around 10%, the total sample size of the trial would will be N=210 patients.

Number of centres 7 centres are included. Research period

* Inclusion period : 60 months
* Treatment period : 6 weeks
* Follow up period : 18 weeks Total research period: 66 months.

Statistical analysis Descriptive Statistics

All study variables will be presented by treatment and overall, by using the appropriate descriptive statistics according to the variable nature, unless otherwise specified:

* Continuous variables: number of non-missing observations, mean, standard deviation, standard error of the mean, minimum, median, maximum.
* Categorical variables: number of non-missing observations and column percentages (N, %) in each category.

Primary efficacy endpoint Primary endpoint: Changes from baseline of IBSSS at V4, will be analyzed by mixed model of ANCOVA with patient as random factor. Baseline value of the score as well as variables a priori known to affect the score will be included in the model.

Secondary efficacy endpoints

* Secondary efficacy variables with binary outcome (i.e. responder status) will be analysed using a Chi-square or Fisher's exact test in a 2 x 2 contingency table to compare active treatment group with placebo. A two-sided overall significance level of 5 % will be used.
* Secondary efficacy variables with continuous variables (i.e. "change from baseline") will be evaluated through an analysis of covariance (ANCOVA) models with fixed effect terms for treatment group and the patient's corresponding baseline value of the parameter as a covariate. The rebound effect will be evaluated with pairwise t-test.

  * Exploratory efficacy endpoints and safety endpoints will be analysed only by descriptive statistics.

For the efficacy endpoints, the following subgroup-analyses will be presented:

* Age (<65 years vs. ≥65 years).
* Baseline abdominal pain severity (pain intensity on the 11-point NRS) <5, ≥5 to <8, ≥8).
* Baseline IBS-SSS score (mild IBS: <175 score points, moderate IBS: 175 to <300 score points, severe IBS: ≥300 score points).
* BMI (<30 kg/m² vs. BMI ≥30 kg/m²).
* Osteopath effect: analysis of data according to the osteopath that practiced the manipulative treatment.
* Analysis according to the subtype of IBS (IBS with constipation, IBS with diarrhoea, Mixed IBS, Unspecified IBS).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes ≥18 years.
* Patient suffering from IBS according to the Rome III criteria:
* IBS SSS must be ≥ 175 at inclusion. Patients who received over the past 5 years a colonoscopy.
* Physical examination without clinically relevant abnormalities during the Screening period.
* Patient is willing to be compliant with study procedures.
* Patient who signed the informed consent before carrying out any procedure related to the study.
* Mentally competent, able to give written informed consent prior to any study-related procedure and compliant to undergo all visits and procedures scheduled in the study
* Medical Insurance

Exclusion Criteria:

* Patient has had surgery that meets any of the following criteria:
* Patient has any elective major surgery planned or expected at any time during the study.
* Use of new drugs indicated in treatment the IBS
* Patient has a history of inflammatory bowel diseases, complicated diverticulosis (i.e. diverticulitis), ischaemic colitis, microscopic colitis.
* Patient has a history of organic abnormalities of the GI tract, intestinal: obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, adhesions or impaired intestinal circulation (e.g., aorto-iliac disease).
* Patient has a history of pancreatitis of any etiology, cholecystitis or of symptomatic gallbladder stone disease in the previous 6 months.
* Patient has an active biliary duct disease or a history of Sphincter of Oddi dysfunction.
* Patient has a history of gluten enteropathy.
* Patient has a history of lactose intolerance as assessed by response to diet.
* Patient has a small intestinal bacterial overgrowth.
* Patient has a current or previous diagnosis of neoplasia (except non-GI neoplasia in complete remission ≥5 years, squamous and basal cell carcinomas and cervical carcinoma in situ).
* Patient has a history of ectopic endometriosis.
* Patient has a history of positive tests for ova or parasites, or clostridium difficile toxin or occult blood in the stool in the previous 6 months.
* Patient has a history of human immunodeficiency virus infection.
* Patient has insulin-dependent diabetes mellitus.
* Patient has a major psychiatric or neurological disorder.
* Patient has an unstable medical condition, which may compromise the efficacy and safety assessments as required in the study and/or require change in concomitant medication.
* Patient has a history of abnormal thyroid function. Patient is candidate for the study if thyroid hormone replacement therapy is stable from at least 2 months.
* Patient has evidence of anemia as confirmed by hemoglobin <9 g/dl during the Screening period.
* Relevant changes in dietary habits, lifestyle, or exercise regimen in the previous 2 months. (dietary habits, lifestyle and exercise regimen should be maintained for the duration of the study).
* Use of prohibited concurrent medication within the previous month
* Pregnancy.
* Patient is not able to understand or collaborate throughout the study.
* Patient has any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the requirements of the study.
* Concomitant participation in a biomedical research trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of IBSSS at V4. | 8 weeks after the first osteopathic manipulative treatment
  It measured by the IBS severity score (IBSSS) after osteopathic manipulative treatment. The IBS Severity Scoring System is a validated measure to assess the severity of IBS symptoms, and can help monitor response to treatment.

SECONDARY OUTCOMES:
Clinical improvement (IBSSS) | 3 and 6 months after the first osteopathic manipulative treatment
  This endpoint will be assessed by the variation of the IBS-SSS during the follow-up period (V5 and V6).
Percentage of patients with improvement at V4, V5 and V6. | 2, 3 and 6 months after the first osteopathic manipulative treatment
  The improvement will be assessed by the reduction of at least of 50 points of the severity of the IBS defined by the IBS -symptom severity score.
Cardinal signs of IBS measured by visual analogic scales | 2, 3 and 6 months after the first osteopathic manipulative treatment
  Cardinal signs of IBS measured by visual analogic scales:
  Constipation, diarrhea, abdominal distension, abdominal pain.
Shape of the stool | 2, 3 and 6 months after the first osteopathic manipulative treatment
  Measured by the Bristol stool form scale
Changes of the severity of IBS | 2, 3 and 6 months after the first osteopathic manipulative treatment
  Changes of the severity of IBS as defined by IBS-SSS.
Depression and anxiety quantified using the Beck Depression Inventory II(BDI-II) questionnaires. | 2, 3 and 6 months after the first osteopathic manipulative treatment
  The intensity of depression is quantified by using the second version of the Beck. Anxiety is scored according to the trait and state questionnaire.
Quality of life defined by IBS-QOL. | 2, 3 and 6 months after the first osteopathic manipulative treatment
  The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment.
Depression and anxiety quantified using the STAI questionnaires. | 2, 3 and 6 months after the first osteopathic manipulative treatment
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bouchoucha, MD, Principal Investigator — Hospital Avicenne
Locations (1):
- Avicenne Hospital, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hundscheid HW, Pepels MJ, Engels LG, Loffeld RJ. Treatment of irritable bowel syndrome with osteopathy: results of a randomized controlled pilot study. J Gastroenterol Hepatol. 2007 Sep;22(9):1394-8. doi: 10.1111/j.1440-1746.2006.04741.x. PMID 17716344
- [Background] Florance BM, Frin G, Dainese R, Nebot-Vivinus MH, Marine Barjoan E, Marjoux S, Laurens JP, Payrouse JL, Hebuterne X, Piche T. Osteopathy improves the severity of irritable bowel syndrome: a pilot randomized sham-controlled study. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):944-9. doi: 10.1097/MEG.0b013e3283543eb7. PMID 22546751
- [Background] Attali TV, Bouchoucha M, Benamouzig R. Treatment of refractory irritable bowel syndrome with visceral osteopathy: short-term and long-term results of a randomized trial. J Dig Dis. 2013 Dec;14(12):654-61. doi: 10.1111/1751-2980.12098. PMID 23981319
- [Background] Muller A, Franke H, Resch KL, Fryer G. Effectiveness of osteopathic manipulative therapy for managing symptoms of irritable bowel syndrome: a systematic review. J Am Osteopath Assoc. 2014 Jun;114(6):470-9. doi: 10.7556/jaoa.2014.098. PMID 24917634
- [Background] Piche T, Pishvaie D, Tirouvaziam D, Filippi J, Dainese R, Tonohouhan M, DeGalleani L, Nebot-Vivinus MH, Payrouse JL, Hebuterne X. Osteopathy decreases the severity of IBS-like symptoms associated with Crohn's disease in patients in remission. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1392-8. doi: 10.1097/MEG.0000000000000219. PMID 25357218